CLINICAL TRIAL: NCT04294394
Title: Rhomboid Block Versus Erector Spinae Block in Thoracotomy
Brief Title: Rhomboid Block,erectör Spiane Block, Thoracotomy
Status: Completed | Type: Observational
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Tahsin Şimşek, medical doctor, Kocaeli Derince Education and Research Hospital
Other Study IDs: 2019/514/150/22
Record Dates: First submitted 2020-03-01; First posted 2020-03-04 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Anesthesia
Keywords: rhomboid block; erectör spinae block

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- rhomboid block: With a 6-13 Mhz linear USG probe, at the thoracal level of 6-7 vertebra in the sagittal position, in the cranio-caudal direction with a 22 G and 100 mm block needle in the medial of the scapula, after entering the facial plane between the rhomboid muscle and the intercostal muscle, 0.25% bupivacaine 20 ml of the local anesthetic solution will be given.
  Interventions: Other: rhomboid block
- erector spinae group: After the patient is taken in the lateral position, the probe T5 is 3 cm lateral to the spinous process, 22 G and 100 mm block needle with 6-13 Mhz linear ultrasonography and the facial plane between the transverse proces and the erector spina muscle is entered, and 20 ml of a local anesthetic solution consisting of 0.25% bupivacaine will be given.
  Interventions: Other: erector spinae block
- control group: For postoperative analgesia, all patients (including Rhomboid block and Erector spinae block) will be administered 100 mg tramadol and 1 gr paracetamol. No additional intervention other than this medical approach will be applied in the control group.
  Interventions: Other: control

INTERVENTIONS:
Other: rhomboid block — Rhombid block, on the other hand, is a method which make up analgesia by providing lokal anestethetic enjection between intercostal muscles and rhomboid muscles and blocks between t3- t9 levels
  Groups: rhomboid block
Other: erector spinae block — The Erector spinae plan block is a recently developed regional block method .Adminestering of lokal anesthetic between the transver proces and erector spinae muscles provides the dorsal and ventral branch blokades of regional spinal nerve and make up the analgesia.İt have a wide range usage such as surgery of thoracal and abdominal area
  Groups: erector spinae group
Other: control — For postoperative analgesia, all patients (including Rhomboid block and Erector spinae block) will be administered 100 mg tramadol and 1 gr paracetamol. No additional intervention other than this medical approach will be applied in the control group.
  Groups: control group

SUMMARY:
Effective analgesia is very important in terms of preventing respiratory, thromboembolic complications and providing early mobilization after open thoracotomy.

Although thoracic epidural analgesia is gold standart method for this aim, it causes common side effects such as hypotension, dural puncture,motor block In recent years, with the effective use of ultrasonography, different regional anesthesia methods have been developed to prevent such complications

DETAILED DESCRIPTION:
A total of 75 patients will be included in the study in three groups: group ESPB, group RIB and control group (group K). Under general anesthesia, patients who will undergo both ESPB and RIB will be applied block with a 22 G and 100 mm block needle, accompanied by ultrasonography, and 20 ml 0.25% bupivacaine. Apart from the standard peroperative analgesia protocol applied to all three groups, no additional procedure will be performed in group control. Postoperative analgesic consumption amount, first analgesic requirement time and visual analog scale (VAS) values of the patients will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-75 years old
* ASA1,2,3 group patients
* Patients undergoing thoracotomy under general anesthesia

Exclusion Criteria:

* The patient's refusal to participate in the study
* Allergy to local anesthetics

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 18 to 75 years old patients will including in this study. Patients Asa Scores shold be ASA1,2,3
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
rhomboid block versus erector spinae block in thorachotomy | the study will comlete in three month
  In this study, we aimed to compare the effects of rhomboid block and erector spinae block in pain control after thoracotomy

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Derince Eğitim Ve Araştırma Hastanesi, Kocaeli, Derince
  - Tahsin Şimşek, Istanbul